CLINICAL TRIAL: NCT00303186
Title: An Observational Study to Evaluate the Cost of the Treatments of the Refractory Psoriatic Arthritis to the Conventional Therapy
Brief Title: Study Evaluating the Cost of the Treatments of the Refractory Psoriatic Arthritis to the Conventional Therapy
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 0881A-101750; B1801109
Record Dates: First submitted 2006-03-14; First posted 2006-03-15 (Estimated); Results first posted 2012-07-30 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-06

CONDITIONS: Arthritis, Psoriatic, Psoriasis
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis; Psoriasis; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to conduct an economic analysis on the cost of conventional therapy as compared to biologic therapy and the direct/indirect costs of disease management in patients with refractory psoriatic arthritis (PsA). Primary outcomes are to qualify the economic burden of refractory PsA care. The secondary outcomes are to assess efficacy, safety, and cost effectiveness of different therapies.

ELIGIBILITY:
Inclusion Criteria:

* Eighteen years of age or older
* Inflammatory arthropathy associated with psoriasis meet the ACR criteria for PsA
* Patients with diagnosis of active and progressive PsA who have failure with conventional treatments

Exclusion Criteria:

* Significant concurrent medical diseases including cancer or a history of cancer, uncontrolled congestive heart failure, myocardial infarctions within 12 months or other clinically significant cardiovascular diseases, immunodeficiency syndromes or concomitant infectious diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with PsA who are failure to the conventional treatments according to the local recommendations, will be enrolled in the study through tertiary referrals centers (HRCs i.e., Hospital Rheumatolgic Centers).
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2005-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- Italy (9):
  - Pfizer Investigational Site, Cagliari, Cagliari
  - Pfizer Investigational Site, Napoli, Campania
  - Pfizer Investigational Site, Prato, FI - Italy
  - Pfizer Investigational Site, Florence, Italy
  - Pfizer Investigational Site, Padua, Padova
  - Pfizer Investigational Site, Potenza, Potenza
  - Pfizer Investigational Site, Reggio Emilia, Reggio Emilia
  - Pfizer Investigational Site, Roma, Roma
  - Pfizer Investigational Site, Benevento

REFERENCES:
- [Derived] Olivieri I, Cortesi PA, de Portu S, Salvarani C, Cauli A, Lubrano E, Spadaro A, Cantini F, Ciampichini R, Cutro MS, Mathieu A, Matucci-Cerinic M, Punzi L, Scarpa R, Mantovani LG; PACE Working Group. Long-term costs and outcomes in psoriatic arthritis patients not responding to conventional therapy treated with tumour necrosis factor inhibitors: the extension of the Psoriatic Arthritis Cost Evaluation (PACE) study. Clin Exp Rheumatol. 2016 Jan-Feb;34(1):68-75. Epub 2015 Dec 3. PMID 26633622
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0881A-101750&StudyName=Study%20Evaluating%20the%20Cost%20of%20the%20Treatments%20of%20the%20Refractory%20Psoriatic%20Arthritis%20to%20the%20Conventional%20Therapy

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: Participants with psoriatic arthritis (PsA) prescribed with tumor necrosis factor (TNF) inhibitors (etanercept, infliximab, adalimumab) for the treatment of refractory PsA to the conventional treatments according to the Italian recommendations of Italian Society of Rheumatology were observed for 60 months.
Period: Overall Study
Arm/Group | All Participants
Started | 107
Completed | 55
Not Completed | 52
Not completed — Other | 52

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 107
Age Continuous [Mean (Standard Deviation); unit: years] | 49.68 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 51
Mean Cost per Participant per Month [Mean (Standard Deviation); unit: Euro/participant-month] — Overall cost was evaluated to quantify burden of Refractory PsA and its treatment, resources absorbed by disease and its care into monetary terms. Overall cost = sum of direct costs (pharmacological treatment; hospitalizations; diagnostic examinations, laboratory analysis and specialist visits; transports) and indirect costs (productivity losses).
  Euro/participant-month
    Overall | 253.20 (324.19)
    Pharmacological treatment | 105.14 (160.53)
    Hospitalizations | 27.92 (104.56)
    Diagnostic, laboratory, specialist visits | 14.12 (22.70)
    Transports | 9.96 (16.03)
    Indirect costs | 96.05 (260.85)

OUTCOME MEASURES:

1. Primary Outcome: Mean Cost Per Participant Per Month at Month 12
Description: Overall cost per participant per month was evaluated as part of health economics evaluation to quantify burden of Refractory PsA and its treatment, resources absorbed by the disease and its care into monetary terms. Overall cost was defined as sum of direct and indirect costs (productivity losses). Direct costs included cost of following cost variables: pharmacological treatment; hospitalizations; diagnostic examinations, laboratory analysis and specialist visits; transports.
Time Frame: Month 12
Population: Intent-to-Treat (ITT) population included all participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: Euro/participant-month
Arm/Group | All Participants
Number analyzed (Participants) | 107
Euro/participant-month
  Overall | 1026.32 (443.86)
  Pharmacological treatment | 970.14 (445.87)
  Hospitalizations | 4.14 (35.46)
  Diagnostic, laboratory, specialist visits | 13.60 (8.96)
  Transports | 11.32 (24.19)
  Indirect costs | 27.11 (52.35)

2. Primary Outcome: Mean Cost Per Participant Per Month at Month 60
Description: as for outcome 1
Time Frame: Month 60
Population: ITT population included all participants who received at least 1 dose of the study medication. Here, 'N' (number of participants analyzed) is signifying those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: Euro/participant-month
Arm/Group | All Participants
Number analyzed (Participants) | 55
Euro/participant-month
  Overall | 986.34 (469.17)
  Pharmacological treatments | 946.70 (462.71)
  Hospitalizations | 16.97 (36.36)
  Diagnostic, laboratory, specialist visits | 8.55 (8.63)
  Transports | 2.58 (4.87)
  Indirect costs | 11.55 (37.06)

3. Primary Outcome: Incremental Cost-effectiveness Ratio (ICER)
Description: ICER: ratio of the incremental cost of treatment over the incremental effectiveness. Incremental cost = difference in cost between baseline and month 60. Effectiveness was defined as quality adjusted life year (QALY) gained, i.e. difference in Euro Quality of Life 5 Dimension (EQ-5D)- health state profile utility score between baseline and month 60. (EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Total score range -0.594 to 1.000; higher score indicates a better health state.)
Time Frame: Baseline up to Month 60
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: ratio
Arm/Group | All Participants
Number analyzed (Participants) | 53
ratio | 39678.6 [24271.2 to 84692.1]

4. Secondary Outcome: Number of Participants With Assessment in Ankylosing Spondylitis (ASAS) 20 Response
Description: ASAS measures symptomatic improvement in Ankylosing Spondylitis (AS) participants. ASAS = 4 domains: participant global assessment of disease activity, pain, function, inflammation. ASAS 20 = 20% improvement from baseline and an absolute change >= 10 units on a 0-100 scale (0=no disease activity; 100=high disease activity) for >= 3 domains, and no worsening in remaining domain.
Time Frame: Month 6, Month 12, Month 18, Month 24, Month 60
Population: ITT population included all participants who received at least 1 dose of the study medication. Here, 'n' is signifying those participants who were evaluated for this measure at the given time points.
Measure: Number; unit: participants
Arm/Group | All Participants
Number analyzed (Participants) | 107
participants
  Month 12 (n=103) | 75
  Month 60 (n=51) | 37

5. Secondary Outcome: Number of Participants Achieving Psoriatic Arthritis Response Criteria (PsARC)
Description: PsARC is comprised of 4 clinical improvement criteria: 1 unit (0-5 Likert scale) improvement on the Physician Global Assessment (PGA); 20% (0-100 scale) improvement on the participant assessments; and 30% reduction in the number of tender joints; and 30% reduction in the number of swollen joints. To achieve a clinical response, the participant must improve in 2 of the 4 PsARC criteria, 1 of which has to be the number of tender or swollen joints and none of the 4 scores could worsen.
Time Frame: Month 6, Month 12, Month 18, Month 24, Month 60
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | All Participants
Number analyzed (Participants) | 107
participants
  Month 12 (n=106) | 86
  Month 60 (n=50) | 38

6. Secondary Outcome: Psoriasis Area and Severity Index (PASI)
Description: Combined assessment of lesion severity and area affected into single score. Body was divided into 4 sections: head, arms, trunk, legs. For each section, percent area of skin involved was estimated: 0= 0% to 6= 90-100%. Severity was estimated by clinical signs: erythema, induration, desquamation; scale: 0= none to 4= maximum. Final PASI = sum of severity parameters for each section*area score*weight of section (head: 0.1, arms: 0.2, body: 0.3, legs: 0.4); total possible score range: 0= no disease to 72= maximal disease.
Time Frame: Baseline, Month 6, Month 12, Month 18, Month 24, Month 60
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 107
units on a scale
  Baseline (n=107) | 5.04 (7.29)
  Month 12 (n=93) | 1.29 (1.69)
  Month 60 (n=53) | 2.08 (3.74)
Statistical Analysis 1: Comparison: All Participants; Statistical analysis was carried out between categories, Baseline and Month 12; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 3.75, 95% CI 2-sided [2.40 to 5.10], Standard Deviation 7.03
Statistical Analysis 2: Comparison: All Participants; Statistical analysis was carried out between categories, Baseline and Month 60; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = 3.72, 95% CI 2-sided [1.65 to 5.78], Standard Deviation 7.47
Statistical Analysis 3: Comparison: All Participants; Statistical analysis was carried out between categories, Month 12 and Month 60; Test type: Superiority or Other; p = 0.518, t-test, 2 sided; Mean Difference (Final Values) = -0.37, 95% CI 2-sided [-1.50 to 0.76], Standard Deviation 4.10

7. Secondary Outcome: Bath Ankylosing Spondylitis Functional Index (BASFI)
Description: BASFI is a validated self assessment tool that determines the degree of functional limitation in AS. Utilizing a Visual Analog Scale (VAS) of 0-10 (0 = easy, 10 = impossible), participants answered 10 questions assessing their ability in completing normal daily activities or physically demanding activities. The BASFI score is a sum of the scores of the 10 questions. Total possible score range: 0-100, where higher score referred to higher impairment in the functional ability.
Time Frame: Baseline, Month 6, Month 12, Month 18, Month 24, Month 60
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 107
units on a scale
  Baseline (n=107) | 43.37 (24.49)
  Month 12 (n=107) | 25.65 (22.53)
  Month 60 (n=53) | 22.46 (22.78)
Statistical Analysis 1: Comparison: All Participants; Statistical analysis was carried out between categories, Baseline and Month 12; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 17.72, 95% CI 2-sided [12.38 to 23.07], Standard Deviation 27.89
Statistical Analysis 2: Comparison: All Participants; Statistical analysis was carried out between categories, Baseline and Month 60; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 12.60, 95% CI 2-sided [6.99 to 18.21], Standard Deviation 20.36
Statistical Analysis 3: Comparison: All Participants; Statistical analysis was carried out between categories, Month 12 and Month 60; Test type: Superiority or Other; p = 0.833, t-test, 2 sided; Mean Difference (Final Values) = -0.55, 95% CI 2-sided [-5.70 to 4.61], Standard Deviation 18.70

8. Secondary Outcome: Bath Ankylosing Spondylitis Disease Activity Index (BASDAI)
Description: BASDAI is a validated self assessment tool used to determine disease activity in participant with Ankylosing Spondylitis (AS). Utilizing a VAS of 0-10 (0=none and 10=very severe) participant's answered 6 questions measuring discomfort, pain and fatigue. The final BASDAI score averages the individual assessments for a final score range of 0-10.
Time Frame: Baseline, Month 6, Month 12, Month 18, Month 24, Month 60
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 107
units on a scale
  Baseline (n=107) | 5.95 (1.82)
  Month 12 (n=107) | 3.23 (2.32)
  Month 60 (n=55) | 3.34 (2.46)
Statistical Analysis 1: Comparison: All Participants; Statistical analysis was carried out between categories, Baseline and Month 12; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 2.72, 95% CI 2-sided [2.26 to 3.18], Standard Deviation 2.39
Statistical Analysis 2: Comparison: All Participants; Statistical analysis was carried out between categories, Baseline and Month 60; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 2.23, 95% CI 2-sided [1.59 to 2.87], Standard Deviation 2.36
Statistical Analysis 3: Comparison: All Participants; Statistical analysis was carried out between categories, Month 12 and Month 60; Test type: Superiority or Other; p = 0.309, t-test, 2 sided; Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-0.83 to 0.27], Standard Deviation 2.03

9. Secondary Outcome: Bath Ankylosing Spondylitis Radiology Index (BASRI)
Description: BASRI- Radiographs of participants with AS were scored using the New York criteria for the sacroiliac joints on a scale of 2 to 4, the lumbar and cervical spine on a scale of 0 to 4 (0 = normal, 1 = suspicious, 2 = mild, 3 = moderate, 4 = severe). These 3 scores were added together to produce the BASRI-spine (BASRI-s) score (range 2 to 12). Similarly, hip joints were scored on a scale of 0 to 4 to give BASRI-hip (BASRI-h). Sum of BASRI-s and BASRI-h produced BASRI-total (BASRI-t) score; total range 2 to 16, higher score represented worse health state.
Time Frame: Baseline, Month 6, Month 12, Month 18, Month 24, Month 60
Population: Data was not statistically analyzed because of insufficient data collected and small sample size achieved.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 0

10. Secondary Outcome: Modified Schober's Test
Description: Measurement in centimeters (cm) of the distance between marks originally placed while the participant was standing erect 10 cm above and 5 cm below the midpoint of a line that joints the posterior superior iliac spines. Distance between marks was re-measured with participant maximally bend forward, knees fully extended, with spine in full flexion.
Time Frame: Baseline, Month 6, Month 12, Month 18, Month 24, Month 60
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | All Participants
Number analyzed (Participants) | 107
cm
  Baseline (n=52) | 10.65 (12.45)
  Month 12 (n=0) | NA (NA) — Data was not analyzed because none of the participants was evaluable for this measure at Month 12.
  Month 60 (n=53) | 5.91 (5.91)
Statistical Analysis 1: Comparison: All Participants; Statistical analysis was carried out between categories, Baseline and Month 60; Test type: Superiority or Other; p = 0.004, t-test, 2 sided; Mean Difference (Final Values) = 1.66, 95% CI 2-sided [1.619 to 8.301], Standard Deviation 11.75

11. Secondary Outcome: Chest Expansion Measurement
Description: Chest expansion, measured in cm, is defined as the difference in thoracic circumference during full expiration versus full inspiration, measured at the fourth intercostal space (nipple line).
Time Frame: Baseline, Month 6, Month 12, Month 18, Month 24, Month 60
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | All Participants
Number analyzed (Participants) | 107
cm
  Baseline (n=52) | 4.38 (5.52)
  Month 12 (n=0) | NA (NA) — Data was not analyzed because none of the participants was evaluable for this measure at Month 12.
  Month 60 (n=52) | 10.85 (16.72)
Statistical Analysis 1: Comparison: All Participants; Statistical analysis was carried out between categories, Baseline and Month 60; Test type: Superiority or Other; p = 0.015, t-test, 2 sided; Mean Difference (Final Values) = -6.76, 95% CI 2-sided [-12.155 to -1.355], Standard Deviation 18.80

12. Secondary Outcome: Occiput-to-wall Distance
Description: Occiput-to-wall distance: distance between the occiput (posterior or back portion of the head) and the wall when the participant stood with heels and shoulder against the wall and the back straight.
Time Frame: Baseline, Month 6, Month 12, Month 18, Month 24, Month 60
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | All Participants
Number analyzed (Participants) | 107
cm
  Baseline (n=51) | 7.02 (6.24)
  Month 12 (n=0) | NA (NA) — Data was not analyzed because none of the participants was evaluable for this measure at Month 12.
  Month 60 (n=54) | 6.24 (5.50)
Statistical Analysis 1: Comparison: All Participants; Statistical analysis was carried out between categories, Baseline and Month 60; Test type: Superiority or Other; p = 0.676, t-test, 2 sided; Mean Difference (Final Values) = 0.44, 95% CI 2-sided [-1.666 to 2.546], Standard Deviation 7.41

13. Secondary Outcome: Maastricht Ankylosing Spondylitis Enthesis Score (MASES)
Description: Assessment of enthesitis was performed in the following 7 domains: 1) 1st costochondral joint left and right, 2) 7th costochondral joint left and right, 3) posterior superior iliac spine left and right, 4) anterior superior iliac spine left and right, 5) iliac crest left and right, 6) 5th lumbar spinous process and 7) proximal insertion of Achilles tendon left and right. Each domain was graded for the presence (1) and absence (0) of tenderness yielding total MASES ranging from 0 (no tenderness) to 13 (worst possible score; severe tenderness).
Time Frame: Baseline, Month 6, Month 12, Month 18, Month 24, Month 60
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 107
units on a scale
  Baseline (n=107) | 3.65 (3.76)
  Month 12 (n=107) | 2.17 (3.52)
  Month 60 (n=54) | 1.43 (2.53)
Statistical Analysis 1: Comparison: All Participants; Statistical analysis was carried out between categories, Baseline and Month 12; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 1.486, 95% CI 2-sided [0.918 to 2.05], Standard Deviation 2.96
Statistical Analysis 2: Comparison: All Participants; Statistical analysis was carried out between categories, Baseline and Month 60; Test type: Superiority or Other; p < 0.001, t-test, 1 sided; Mean Difference (Final Values) = 2.00, 95% CI 2-sided [1.01 to 2.99], Standard Deviation 3.64
Statistical Analysis 3: Comparison: All Participants; Statistical analysis was carried out between categories, Month 12 and Month 60; Test type: Superiority or Other; p = 0.223, t-test, 2 sided; Mean Difference (Final Values) = 0.56, 95% CI 2-sided [-0.35 to 1.46], Standard Deviation 3.32

14. Secondary Outcome: Number of Swollen and Tender Joints
Description: Number of swollen joints was determined by examination of 66 joints and identifying when swelling was present. The number of swollen joints was recorded on the joint assessment form at each visit, no swelling = 0, swelling =1. Number of tender joints was determined by examining 68 joints and identified the joints that were painful under pressure or to passive motion. The number of tender joints was recorded on the joint assessment form at each visit, no tenderness = 0, tenderness = 1.
Time Frame: Baseline, Month 6, Month 12, Month 18, Month 24, Month 60
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | All Participants
Number analyzed (Participants) | 107
joints
  Baseline: swollen joints (n=107) | 7.60 (6.39)
  Baseline: tender joints (n=107) | 16.97 (11.8)
  Month 12: swollen joints (n=107) | 1.26 (2.54)
  Month 12: tender joints (n=107) | 7.97 (10.18)
  Month 60: swollen joints (n=55) | 0.96 (1.94)
  Month 60: tender joints (n=55) | 5.49 (9.34)
Statistical Analysis 1: Comparison: All Participants; Statistical analysis was carried out between categories, Baseline: swollen joints and Month 12: swollen joints; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 6.33, 95% CI 2-sided [5.10 to 7.47], Standard Deviation 5.94
Statistical Analysis 2: Comparison: All Participants; Statistical analysis was carried out between categories, Baseline: swollen joints and Month 60: swollen joints; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 6.20, 95% CI 2-sided [4.48 to 7.92], Standard Deviation 6.35
Statistical Analysis 3: Comparison: All Participants; Statistical analysis was carried out between categories, Month 12: swollen joints and Month 60: swollen joints; Test type: Superiority or Other; p = 0.479, t-test, 2 sided; Mean Difference (Final Values) = 0.20, 95% CI 2-sided [-0.36 to 0.76], Standard Deviation 2.09
Statistical Analysis 4: Comparison: All Participants; Statistical analysis was carried out between categories, Baseline: tender joints and Month 12: tender joints; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided; Mean Difference (Final Values) = 9.00, 95% CI 2-sided [6.86 to 11.13], Standard Deviation 11.16
Statistical Analysis 5: Comparison: All Participants; Statistical analysis was carried out between categories, Baseline: tender joints and Month 60: tender joints; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 8.60, 95% CI 2-sided [6.10 to 11.10], Standard Deviation 9.25
Statistical Analysis 6: Comparison: All Participants; Statistical analysis was carried out between categories, Month 12: tender joints and Month 60: tender joints; Test type: Superiority or Other; p = 0.588, t-test, 2 sided; Mean Difference (Final Values) = 0.66, 95% CI 2-sided [-1.76 to 3.07], Standard Deviation 8.92

15. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 20% (ACR20) Response
Description: ACR20 response: greater than or equal to (>=) 20 percent (%) improvement in tender joint count; >= 20% improvement in swollen joint count; and >= 20% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and C-Reactive Protein (CRP).
Time Frame: Month 6, Month 12, Month 18, Month 24, Month 60
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 107
percentage of participants
  Month 12 (n=107) | 62.6
  Month 60 (n=51) | 70.6

16. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 50% (ACR50) Response
Description: ACR50 response: >= 50% improvement in tender joint count; >= 50% improvement in swollen joint count; and >= 50% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the HAQ); and CRP.
Time Frame: Month 6, Month 12, Month 18, Month 24, Month 60
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 107
percentage of participants
  Month 12 (n=106) | 41.5
  Month 60 (n=51) | 43.1

17. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 70% (ACR70) Response
Description: ACR70 response: >= 70% improvement in tender joint count; >= 70% improvement in swollen joint count; and >= 70% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the HAQ); and CRP.
Time Frame: Month 6, Month 12, Month 18, Month 24, Month 60
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 107
percentage of participants
  Month 12 (n=106) | 19.8
  Month 60 (n=52) | 26.9

18. Secondary Outcome: Radiographic Score Based on Wassenberg
Description: Radiographic score based on wassenberg consisted of 2 sub-scores, proliferation score (PS) assessing bone proliferation and destruction score (DS) assessing joint surface destruction. Score range for PS and DS was 0 to 160 (where higher score represented higher bone proliferation) and 0 to 200 (where higher score represented higher destruction), respectively. Total score = sum of PS and DS (range 0 to 360); higher score represented worse state.
Time Frame: Baseline, Month 12, Month 24, Month 60
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 107
units on a scale
  Baseline (n=77) | 13.58 (24.21)
  Month 12 (n=96) | 11.66 (21.37)
  Month 60 (n=14) | 28.29 (32.93)
Statistical Analysis 1: Comparison: All Participants; Statistical analysis was carried out between categories, Baseline and Month 12; Test type: Superiority or Other; p = 0.330, t-test, 2 sided; Mean Difference (Final Values) = 1.26, 95% CI 2-sided [-1.30 to 3.82], Standard Deviation 11.29
Statistical Analysis 2: Comparison: All Participants; Statistical analysis was carried out between categories, Baseline and Month 60; Test type: Superiority or Other; p = 0.449, t-test, 2 sided; Mean Difference (Final Values) = -8.56, 95% CI 2-sided [-33.37 to 16.26], Standard Deviation 32.28
Statistical Analysis 3: Comparison: All Participants; Statistical analysis was carried out between categories, Month 12 and Month 60; Test type: Superiority or Other; p = 0.165, t-test, 2 sided; Mean Difference (Final Values) = -15.00, 95% CI 2-sided [-37.04 to 7.04], Standard Deviation 38.17

19. Secondary Outcome: Patient Global Assessment (PtGA) of Disease Activity Score
Description: Measured using a 100 millimeter (mm) VAS ranging from 0 mm = very good to 100 mm = very bad.
Time Frame: Baseline, Month 6, Month 12, Month 18, Month 24, Month 60
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | All Participants
Number analyzed (Participants) | 107
mm
  Baseline (n=107) | 63.51 (17.25)
  Month 12 (n=107) | 32.07 (22.33)
  Month 60 (n=55) | 33.16 (24.50)
Statistical Analysis 1: Comparison: All Participants; Statistical analysis was carried out between categories, Baseline and Month 12; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 31.18, 95% CI 2-sided [26.44 to 35.91], Standard Deviation 24.48
Statistical Analysis 2: Comparison: All Participants; Statistical analysis was carried out between categories, Baseline and Month 60; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 28.76, 95% CI 2-sided [22.42 to 35.10], Standard Deviation 23.24
Statistical Analysis 3: Comparison: All Participants; Statistical analysis was carried out between categories, Month 12 and Month 60; Test type: Superiority or Other; p = 0.538, t-test, 2 sided; Mean Difference (Final Values) = -2.05, 95% CI 2-sided [-8.70 to 4.60], Standard Deviation 24.60

20. Secondary Outcome: Physician Global Assessment (PGA) of Disease Activity
Description: Physician Global Assessment of Disease Activity was measured on a 0 to 100 mm VAS, with 0 mm = no disease activity.
Time Frame: Baseline, Month 6, Month 12, Month 18, Month 24, Month 60
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | All Participants
Number analyzed (Participants) | 107
mm
  Baseline (n=107) | 60.15 (13.33)
  Month 12 (n=107) | 26.43 (18.53)
  Month 60 (n=50) | 23.00 (16.42)
Statistical Analysis 1: Comparison: All Participants; Statistical analysis was carried out between categories, Baseline and Month 12; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 33.83, 95% CI 2-sided [30.04 to 37.63], Standard Deviation 19.60
Statistical Analysis 2: Comparison: All Participants; Statistical analysis was carried out between categories, Baseline and Month 60; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 38.04, 95% CI 2-sided [31.96 to 44.12], Standard Deviation 21.17
Statistical Analysis 3: Comparison: All Participants; Statistical analysis was carried out between categories, Month 12 and Month 60; Test type: Superiority or Other; p = 0.343, t-test, 2 sided; Mean Difference (Final Values) = 2.38, 95% CI 2-sided [-2.62 to 7.38], Standard Deviation 17.59

21. Secondary Outcome: Visual Analogue Scale for Pain (VAS-pain)
Description: 100 mm line (VAS) marked by participant. Intensity of pain range (over past week): 0 = no pain to 100 = worst possible pain.
Time Frame: Baseline, Month 6, Month 12, Month 18, Month 24, Month 60
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | All Participants
Number analyzed (Participants) | 107
mm
  Baseline (n=107) | 62.83 (21.10)
  Month 12 (n=107) | 31.39 (23.59)
  Month 60 (n=51) | 31.92 (26.51)
Statistical Analysis 1: Comparison: All Participants; Statistical analysis was carried out between categories, Baseline and Month 12; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 31.18, 95% CI 2-sided [25.88 to 36.49], Standard Deviation 27.56
Statistical Analysis 2: Comparison: All Participants; Statistical analysis was carried out between categories, Baseline and Month 60; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 28.80, 95% CI 2-sided [21.52 to 36.09], Standard Deviation 25.89
Statistical Analysis 3: Comparison: All Participants; Statistical analysis was carried out between categories, Month 12 and Month 60; Test type: Superiority or Other; p = 0.301, t-test, 2 sided; Mean Difference (Final Values) = -3.33, 95% CI 2-sided [-9.74 to 3.07], Standard Deviation 22.77

22. Secondary Outcome: Erythrocyte Sedimentation Rate (ESR)
Description: ESR is a laboratory test that provides a non-specific measure of inflammation. The test assesses the rate at which red blood cells fall in a test tube. Normal range is 0-30 millimeter/hour (mm/hr). A higher rate is consistent with inflammation.
Time Frame: Baseline, Month 6, Month 12, Month 18, Month 24, Month 60
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | All Participants
Number analyzed (Participants) | 107
mm/hr
  Baseline (n=105) | 42.07 (121.18)
  Month 12 (n=104) | 16.36 (16.79)
  Month 60 (n=49) | 16.61 (14.77)
Statistical Analysis 1: Comparison: All Participants; Statistical analysis was carried out between categories, Baseline and Month 12; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 26.21, 95% CI 2-sided [2.01 to 50.40], Standard Deviation 123.20
Statistical Analysis 2: Comparison: All Participants; Statistical analysis was carried out between categories, Baseline and Month 60; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 13.19, 95% CI 2-sided [7.81 to 18.57], Standard Deviation 18.30
Statistical Analysis 3: Comparison: All Participants; Statistical analysis was carried out between categories, Month 12 and Month 60; Test type: Superiority or Other; p = 0.132, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -2.31, 95% CI 2-sided [-6.40 to 1.77], Standard Deviation 14.07

23. Secondary Outcome: C-reactive Protein (CRP)
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement.
Time Frame: Baseline, Month 6, Month 12, Month 18, Month 24, Month 60
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: milligram/deciliter (mg/dL)
Arm/Group | All Participants
Number analyzed (Participants) | 107
milligram/deciliter (mg/dL)
  Baseline (n=104) | 59.41 (148.83)
  Month 12 (n=103) | 42.07 (129.70)
  Month 60 (n=46) | 2.30 (3.60)
Statistical Analysis 1: Comparison: All Participants; Statistical analysis was carried out between categories, Baseline and Month 12; Test type: Superiority or Other; p < 0.0005, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 16.26, 95% CI 2-sided [-13.52 to 46.04], Standard Deviation 150.10
Statistical Analysis 2: Comparison: All Participants; Statistical analysis was carried out between categories, Baseline and Month 60; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 52.81, 95% CI 2-sided [22.33 to 83.29], Standard Deviation 100.25
Statistical Analysis 3: Comparison: All Participants; Statistical analysis was carried out between categories, Month 12 and Month 60; Test type: Superiority or Other; p = 0.034, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 33.40, 95% CI 2-sided [-10.84 to 77.64], Standard Deviation 147.25

24. Secondary Outcome: Duration of Morning Stiffness
Description: Duration of morning stiffness is defined as the time elapsed when participant woke up in the morning and was able to resume normal activities without stiffness in minutes (if none was present = 0; if morning stiffness was continuing, average of duration of stiffness over the past 3 days was reported; if stiffness persisted the entire day, 1440 minutes [24 hours*60 minutes] was recorded).
Time Frame: Baseline, Month 6, Month 12, Month 18, Month 24, Month 60
Population: Data was not statistically analyzed because of insufficient data collected and small sample size achieved.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | All Participants
Number analyzed (Participants) | 0

25. Secondary Outcome: Health Assessment Questionnaire (HAQ)
Description: HAQ: participant-reported assessment of ability to perform tasks: 1) dress/groom; 2) arise; 3) eat; 4) walk; 5) reach; 6) grip; 7) hygiene; and 8) common activities over past week. Each item scored on 4-point Likert scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty.
Time Frame: Baseline, Month 6, Month 12, Month 18, Month 24, Month 60
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 107
units on a scale
  Baseline (n=107) | 1.14 (0.57)
  Month 12 (n=93) | 0.71 (0.56)
  Month 60 (n=55) | 0.65 (0.61)
Statistical Analysis 1: Comparison: All Participants; Statistical analysis was carried out between categories, Baseline and Month 12; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 0.48, 95% CI 2-sided [0.35 to 0.62], Standard Deviation 0.66
Statistical Analysis 2: Comparison: All Participants; Statistical analysis was carried out between categories, Baseline and Month 60; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 0.41, 95% CI 2-sided [0.26 to 0.56], Standard Deviation 0.56
Statistical Analysis 3: Comparison: All Participants; Statistical analysis was carried out between categories, Month 12 and Month 60; Test type: Superiority or Other; p = 0.600, t-test, 2 sided; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.24 to 0.14], Standard Deviation 0.61

26. Secondary Outcome: Euro Quality of Life (EQ-5D)- Health State Profile Utility Score
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single utility score. It assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state ("confined to bed"). Scoring formula developed by EuroQol Group assigns a utility value for each domain in the profile. Score is transformed and results in a total score range -0.594 to 1.000; higher score indicates a better health state.
Time Frame: Baseline, Month 6, Month 12, Month 18, Month 24, Month 60
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 107
units on a scale
  Baseline (n=105) | 0.38 (0.32)
  Month 12 (n=107) | 0.63 (0.27)
  Month 60 (n=55) | 0.63 (0.28)
Statistical Analysis 1: Comparison: All Participants; Statistical analysis was carried out between categories, Baseline and Month 12; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 0.25, 95% CI 2-sided [0.18 to 0.30], Standard Deviation 0.31
Statistical Analysis 2: Comparison: All Participants; Statistical analysis was carried out between categories, Baseline and Month 60; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-0.31 to -0.12], Standard Deviation 0.34
Statistical Analysis 3: Comparison: All Participants; Statistical analysis was carried out between categories, Month 12 and Month 60; Test type: Superiority or Other; p = 0.789, t-test, 2 sided; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.08 to 0.06], Standard Deviation 0.27

27. Secondary Outcome: Euro Quality of Life (EQ-5D)- Visual Analog Scale (VAS)
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single index value. The VAS component rates current health state on a scale from 0 mm (worst imaginable health state) to 100 mm (best imaginable health state); higher scores indicate a better health state.
Time Frame: Baseline, Month 6, Month 12, Month 18, Month 24, Month 60
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | All Participants
Number analyzed (Participants) | 107
mm
  Baseline (n=105) | 46.91 (20.98)
  Month 12 (n=107) | 66.76 (20.37)
  Month 60 (n=54) | 64.17 (21.08)
Statistical Analysis 1: Comparison: All Participants; Statistical analysis was carried out between categories, Baseline and Month 12; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 19.40, 95% CI 2-sided [14.59 to 24.22], Standard Deviation 25.00
Statistical Analysis 2: Comparison: All Participants; Statistical analysis was carried out between categories, Baseline and Month 60; Test type: Superiority or Other; p = 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -12.68, 95% CI 2-sided [-18.77 to -6.59], Standard Deviation 22.08
Statistical Analysis 3: Comparison: All Participants; Statistical analysis was carried out between categories, Month 12 and Month 60; Test type: Superiority or Other; p = 0.115, t-test, 2 sided; Mean Difference (Final Values) = 4.85, 95% CI 2-sided [-1.21 to 10.92], Standard Deviation 22.22

28. Secondary Outcome: 36-Item Short-Form Health Survey (SF-36)
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning) and was reported as 2 summary scores; Physical Component Score and Mental Component Score. Total score range for the summary scores = 0-100 where higher scores represented higher level of functioning.
Time Frame: Baseline, Month 6, Month 12, Month 18, Month 24, Month 60
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 107
units on a scale
  Baseline: Physical Component Score (n=94) | 31.88 (8.22)
  Baseline: Mental Component Score (n=94) | 40.80 (6.50)
  Month 12: Physical Component Score (n=103) | 40.44 (12.06)
  Month 12: Mental Component Score (n=103) | 39.15 (8.08)
  Month 60: Physical Component Score (n=55) | 40.77 (9.54)
  Month 60: Mental Component Score (n=55) | 45.03 (12.42)
Statistical Analysis 1: Comparison: All Participants; Statistical analysis was carried out between categories, Baseline: physical component score and Month 12: physical component score; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -7.41, 95% CI 2-sided [-10.34 to -4.47], Standard Deviation 10.10
Statistical Analysis 2: Comparison: All Participants; Statistical analysis was carried out between categories, Baseline: physical component score and Month 60: physical component score; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -5.94, 95% CI 2-sided [-8.56 to -3.32], Standard Deviation 9.13
Statistical Analysis 3: Comparison: All Participants; Statistical analysis was carried out between categories, Month 12: physical component score and Month 60: physical component score; Test type: Superiority or Other; p = 0.308, t-test, 2 sided; Mean Difference (Final Values) = 1.25, 95% CI 2-sided [-1.19 to 3.68], Standard Deviation 8.83
Statistical Analysis 4: Comparison: All Participants; Statistical analysis was carried out between categories, Baseline: mental component score and Month 12: mental component score; Test type: Superiority or Other; p = 0.589, t-test, 2 sided; Mean Difference (Final Values) = -0.67, 95% CI 2-sided [-3.14 to 1.80], Standard Deviation 8.51
Statistical Analysis 5: Comparison: All Participants; Statistical analysis was carried out between categories, Baseline: mental component score and Month 60: mental component score; Test type: Superiority or Other; p = 0.003, t-test, 2 sided; Mean Difference (Final Values) = -5.59, 95% CI 2-sided [-9.12 to -2.06], Standard Deviation 12.29
Statistical Analysis 6: Comparison: All Participants; Statistical analysis was carried out between categories, Month 12: mental component score and Month 60: mental component score; Test type: Superiority or Other; p = 0.002, t-test, 2 sided; Mean Difference (Final Values) = -5.70, 95% CI 2-sided [-9.23 to -2.18], Standard Deviation 12.80

ADVERSE EVENTS:
Time Frame: Year 3 up to Year 5
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/107
Other Adverse Events (participants affected / at risk) | 8/107
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=107)
Abdominal colic (General disorders) | 2
Pyrexia (General disorders) | 2
Benign prostatic hyperplasia (General disorders) | 1
Bronchopneumonia (General disorders) | 1
Epidermal cyst (General disorders) | 1
Gastrointestinal tract adenoma (General disorders) | 1
Hiatus hernia (General disorders) | 1
Osteoarthritis (General disorders) | 1
Psoriasis flare-up (General disorders) | 1
Renal colic (General disorders) | 1
Soft tissues neoplasms benign (General disorders) | 1
Thrombocytopenia (General disorders) | 1
Transaminases increased (General disorders) | 1

LIMITATIONS AND CAVEATS:
Results were not summarized for Month 6, 18 and 24 due to insufficient data collected and small sample size achieved at the time points.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.